CLINICAL TRIAL: NCT01227304
Title: SMOOCH - Small Volume Challenges to Predict Volume Responsiveness: Prospective Interventional Study
Acronym: SMOOCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Wolfgang Huber, Klinikumr rechts der Isar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SMOOCH-1
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Prediction of Volume Responsiveness

ARMS (1):
- Test of volume responsiveness using crystalloids (Experimental)
  Interventions: Device: PiCCO-parameter-guided volume challenge

INTERVENTIONS:
Device: PiCCO-parameter-guided volume challenge — Infusion of 7ml/kg crystalloid over 30 minutes, Performing transpulmonary thermodilutions after 0min, 15min and 30min. Recording of pulse contour cardiac index, heart rate and mean arterial pressure after 5, 10, 15, 20, 25 and 30min. Catecholamines are kept stable over the 30min period.

SUMMARY:
* test for volume responsiveness
* PiCCO-guided infusion over a pre-defined period of time

ELIGIBILITY:
Inclusion Criteria:

* Patients are equipped with PiCCO monitoring independently to the study.
* One criteria of decreased usefulness of the parameters of preload/volume responsiveness available using the PiCCO device:

  1. Femoral access of the central venous catheter precluding application of the normal ranges of global enddiastolic volume index and central venous pressure.
  2. Absence of sinus rhythm and/or controlled ventilation precluding the use of stroke volume variation.
  3. Evidence of increased intraabdominal pressure which is known to further reduce the usefulness of central venous pressure.
  4. Contradictory suggestions by stroke volume variation and global enddiastolic volume index.
  5. Intolerance of passive leg raising.
  6. Absence of therapeutic alternatives to volume resuscitation.

Exclusion Criteria:

* Extravascular volume-over plus: global enddiastolic volume index > 1000ml/sqm
* Pulmonary edema: extravascular lungwater index > 20ml/kg
* Cardiogenic shock without volume deficiency (cardiac index <2L/min; global enddiastolic volume index > 850ml/sqm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-07; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Prediction of volume responsiveness defined as an increase in Cardiac Index of ≥ 15% after transpulmonary thermodilution measurement of 15 minutes | 15 minutes after start of infusion
Prediction of volume responsiveness defined as an increase in Cardiac Index of ≥ 15% after transpulmonary thermodilution measurement of 30 minutes | 30 minutes after start of infusion

SECONDARY OUTCOMES:
Predictive capabilities of Cardiac Index (measured by pulse contour) | within 30 minutes after start of infusion
Comparison of global enddiastolic volume index to baseline values | 30 minutes after start of infusion
Comparison of central venous pressure levels to baseline values | 30 minutes after start of infusion

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Medical Department, Klinikum rechts der Isar, Munich, Germany